CLINICAL TRIAL: NCT05762601
Title: Cellular precOnditioning for Post-Surgical Myocardial Ischemic Complications - Observational Study
Acronym: COSMIC
Status: Recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20220330-01H
Record Dates: First submitted 2023-02-08; First posted 2023-03-09 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Complication; Myocardial Infarction; Myocardial Ischemia; Myocardial Injury
Keywords: Myocardial injury after noncardiac surgery; Perioperative myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Only plasma will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to collect health data on people who are at high risk of having heart complications and are having a surgery that is not on the heart. The main questions it aims to answer are:

* Is this study feasible in terms of recruiting enough people to participate in this study?
* How often do heart complications happen in people who are at high risk of heart complications and are having a surgery that is not on the heart?

Participants will have their usual care and will also be asked to:

* Have extra bloodwork done
* Complete some surveys
* Have two echocardiograms (ultrasounds of the heart)
* Continue to follow-up with the research team for one year after their surgery

Researchers will compare how often heart complications occur in this high risk population to a future study where participants will receive stem cells before their surgery.

DETAILED DESCRIPTION:
This observational trial protocol is to collect baseline health data from participants undergoing intermediate to high-risk surgery and at high risk of developing perioperative myocardial ischemic complications for an upcoming Phase 1 trial that determines the feasibility of intravenous delivery of umbilical cord-derived (UC) mesenchymal stromal cells (MSCs) in the same patient population. Participants enrolled in this protocol, however, will not receive cell product; they will receive standard of care and serve as a lead in control group for the interventional study.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all 5 inclusion criteria to be eligible:

* Referred for elective intermediate to high risk noncardiac surgery as defined by the American Heart Association guidelines (e.g., intrathoracic, open intraabdominal, or open vascular surgery)
* 45 years of age or older
* Revised cardiac risk index ≥ 2
* NT-proBNP level of ≥ 200 pg/mL
* Able to provide informed consent

Exclusion Criteria:

* Experience an acute coronary syndrome, myocardial infarction, heart failure, or stroke within preceding 3 months
* Coronary revascularization anticipated during the study period
* Severe mitral/aortic valve stenosis
* Evidence of clinically significant arrhythmia in last three months.
* Major surgical procedure in previous 3 months
* History of malignancy requiring surgery, chemotherapy, immunotherapy, or radiation within previous 5 years
* Ongoing malignancy requiring surgical resection
* Women who are pregnant, breastfeeding, or of childbearing potential who are unable to use a medically acceptable form of contraception throughout the study
* Received any experimental cell therapy previously
* Unable to provide written informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Ottawa Hospital
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Participant Recruitment | 1 year
  Our primary outcome is the feasibility of participant recruitment. This will be determined by measurements of recruitment efficiency: 1) proportion of potentially eligible participants that are successfully screened; 2) proportion of participants successfully screened who do not enroll (reason for failure to enroll will be recorded).
Baseline Frequency of adverse events and serious adverse events | 1 year
  To determine the baseline frequency of adverse events and serious adverse events in this high risk population

SECONDARY OUTCOMES:
Quality of life of participants | 1 year
  The EQ-5D-5L questionnaire will be used. This questionnaire measures quality of life using five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj M Lalu, MD, PhD, Principal Investigator — The Ottawa Hospital Research Institute, The Ottawa Hospital, University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lalu MM, Mazzarello S, Zlepnig J, Dong YYR, Montroy J, McIntyre L, Devereaux PJ, Stewart DJ, David Mazer C, Barron CC, McIsaac DI, Fergusson DA. Safety and Efficacy of Adult Stem Cell Therapy for Acute Myocardial Infarction and Ischemic Heart Failure (SafeCell Heart): A Systematic Review and Meta-Analysis. Stem Cells Transl Med. 2018 Dec;7(12):857-866. doi: 10.1002/sctm.18-0120. Epub 2018 Sep 26. PMID 30255989